CLINICAL TRIAL: NCT05588544
Title: Effect of Adjunctive YSGG Application in Healing Following Periodontal Treatment
Brief Title: YSGG Application in Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Park, Jung Soo, Clinical assistant professor, Korea University Anam Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019AN0551
Record Dates: First submitted 2022-10-11; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP only (Active Comparator): Periodontal treatment by scaling and root planning
  Interventions: Procedure: Er,Cr:YSGG laser
- SRP + laser (Experimental): Periodontal treatment by Laser-assisted scaling and root planning
  Interventions: Procedure: Er,Cr:YSGG laser

INTERVENTIONS:
Procedure: Er,Cr:YSGG laser — Use of laser at the degranulation step of the treatment

SUMMARY:
Adjunctive use of Er,Cr:YSGG (erbium-chromium-yttrium-scandium-gallium-garnet) laser in combination with conventional, mechanical periodontal treatment may benefit in complete decontamination of the periodontal pocket leading to improved early healing and better long term clinical result. Radial firing periodontal tip (RFPT) offered by the Er,Cr:YSGG system is devised to let irradiation primarily in radial pattern (85%) with lesser portion in straight manner (15%), meaning laser beams are effectively emitted to affected root surface and inner epithelium of periodontal pocket with simple tip management. Therefore, using Er,Cr:YSGG laser with RFPT could be the best option for periodontal laser therapy. The aim of this study is to investigate adjunctive treatment effect using Er,Cr:YSGG laser and RFPT in moderate to severe periodontitis patients. Study subjects are randomly allocated to either 'scaling and root planing (SRP) only' or 'SRP + laser therapy' group. Periodontal parameters including probing pocket depth (PPD), clinical attachment level (CAL), modified gingival index (MGI), and plaque index (PI) are recorded at baseline and 8 weeks after treatment. Gingival crevicular fluid (GCF) samples are obtained using paper strips at baseline, 1w, 2w, 4w, and 8w post op. to determine laser-induced effect in early wound healing. Cytokine levels are evaluated from the GCF samples taken.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of stage III or IV periodontitis based on the 2017 periodontitis classification (Tonetti, Greenwell, & Kornman, 2018);
2. minimum of two teeth with probing depth (PD) ≥ 6 mm and radiographic bone loss in at least two quadrants of the whole dentition;
3. each quadrant with a minimum of four teeth; and
4. systemically healthy patients.

Exclusion Criteria:

1. history of periodontal treatment in the previous six months;
2. antibiotic medication in recent three months;
3. under steroid therapy or taking any anti-inflammatory drugs in recent three months;
4. history of any systemic disease that may influence the periodontal condition and treatment outcome, including diabetes mellitus, cancer, metabolic diseases, cardiovascular disease, and rheumatoid arthritis;
5. pregnancy or breastfeeding; and
6. smoking habits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Change of Modified gingival index | 1, 2, 4, and 8 week post-operatively
  Level of gingival inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Jung Soo Park, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No